CLINICAL TRIAL: NCT00140439
Title: Improving Asthma Outcomes in a High Morbidity Urban Pediatric Population: an Emergency Department-based Randomized Clinical Trial
Brief Title: Improving Asthma Outcomes in an Urban Pediatric Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stephen J. Teach, MD, MPH (Other)
Collaborators: American Academy of Allergy, Asthma, and Immunology (Other); Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor-Investigator, Stephen J. Teach, MD, MPH, MD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: RWJ EDDP
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Asthma
Keywords: asthma; emergency department; compliance; randomized clinical trial
MeSH Terms: conditions — Asthma; Emergencies; Patient Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Emergency Department based asthma follow-up clinic — The clinical activities of the intervention followed a fully specified protocol and provided education and care in three domains:
  1. Asthma self-monitoring and management: Educators first reviewed the basic physiology of asthma with emphasis on its chronicity. After evaluating asthma severity and treatment history, the physician completed an individualized medical action plan (MAP) and provided any necessary device teaching.
  2. Environmental modification and trigger control: After evaluation of potential environmental triggers in the home, each family was educated on their control. Each child was provided hypoallergenic bed encasings.
  3. Linkages and referrals to ongoing primary care: Clinic staff stressed the importance of longitudinal asthma care by a PCP. A full report of the clinic visit was mailed to each child's PCP. In addition, the asthma educator scheduled a follow-up appointment with the PCP within 4 weeks

SUMMARY:
Little is known about how ED-based programs can help to reduce pediatric ED visits for asthma. The current study evaluated a novel intervention in which the ED itself became the site of highly individualized, comprehensive follow-up asthma care. It sought to determine if such an intervention could decrease subsequent unscheduled visits for asthma while improving asthma quality of life.

DETAILED DESCRIPTION:
Prospective, randomized clinical trial of a single visit to a specialized emergency department-based asthma follow-up clinic occurring 2-15 days after emergency department care for an acute exacerbation. All patients were followed for 6 months. Analysis was by intention-to-treat with adjustment for baseline differences. Our primary hypothesis was that this intervention would decrease subsequent unscheduled visits (both to EDs and other sources of urgent care) for asthma over a six-month follow-up period. We further hypothesized that the intervention would decrease hospitalizations for asthma, improve compliance with an individualized medical plan and with trigger control, increase scheduled primary care practitioner (PCP) visits for routine asthma care, and decrease asthma symptoms while improving asthma quality of life (QOL).

ELIGIBILITY:
Inclusion Criteria:

1. age between 12 months and 17 years, inclusive;
2. prior physician-diagnosed asthma;
3. ≥1 other unscheduled visit for asthma in the previous 6 months and/or ≥1 hospitalization for asthma in the prior 12 months;
4. a parent/guardian available for interview;
5. residence in Washington, DC or a contiguous Maryland county; and
6. requirement for ≥3 doses of nebulized albuterol in the ED at the time of enrollment.

Exclusion Criteria:

1. significant medical co-morbidities affecting the cardiorespiratory system;
2. a visit to an allergist or a pulmonologist in the prior 6 months;
3. ≥2 of the following: a current written asthma medical action plan, current use of >1 controller medication, or a scheduled visit for asthma care with their PCP in the prior two weeks;
4. enrollment in another asthma research study;
5. unavailability for telephone follow-up; or
6. primary language other than English or Spanish.

Ages: 12 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 488 (Actual)
Dates: Start 2002-04; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Unscheduled visits for asthma | 6 months following enrollment

SECONDARY OUTCOMES:
Hospitalizations for asthma | 6 months following enrollment
Compliance | 6 months following enrollment
Quality of Life | 6 months following enrollment
Morbidity | 6 months following enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Teach, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States